CLINICAL TRIAL: NCT04767516
Title: Multicenter Registry of Subcutaneous ICD Patients
Brief Title: Multicenter Subcutaneous ICD Registry
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Köln (Other)
Collaborators: Uniklinik Ulm (Unknown); St.Barts Hospital, London (Unknown); VCU Hospital, Richmond (Unknown); University Hospital, Bordeaux (Other); University Hospital Southampton NHS Foundation Trust (Other); Hospital La Fe de Valencia (Unknown); Med.Hochschule Hannover (Unknown); EVKLN Duisburg (Unknown); Veterans Affairs Hospital San Juan (Unknown); Colorado Childrens Hospital (Unknown); Stanford Healthcare (Unknown); Uniklinik Giessen (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21-1128
Record Dates: First submitted 2021-02-11; First posted 2021-02-23 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: ICD; ICD Malfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This multicenter registry aims to collect data regarding S-ICD longevity, and battery and lead failure rates. Only clinically collected data is gathered in this registry.

ELIGIBILITY:
Inclusion Criteria:

* S/P S-ICD Implantation

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an S-ICD
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Generator Explantation | from baseline to incidence of explantation through study completion, an average of 5 year
  Incidence of S-ICD generator explantation, due to battery depletion, infection or system upgrade. Assessed by medical records and device interrogation.
Lead Failure | from baseline to incidence of lead failure,through study completion, an average of 5 year
  Incidence of S-ICD lead failure. Assessed by medical records and device interrogation.

SECONDARY OUTCOMES:
Battery Longevity | from baseline to incidence of battery depletion through study completion, an average of 5 year
  Incidence of regular battery depletion. Assessed by medical records and device interrogation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Luker J, Strik M, Andrade JG, Raymond-Paquin A, Elrefai MH, Roberts PR, Perez OC, Kron J, Koneru J, Franqui-Rivera H, Sultan A, Ernst A, Schmitt J, Pott A, Veltmann C, Srinivasan NT, Collinson J, van Stipdonk AMW, Linz D, Fluschnik N, Tonnis T, Haeberlin A, Ploux S, Steven D. Incidence of premature battery depletion in subcutaneous cardioverter-defibrillator patients: insights from a multicenter registry. J Interv Card Electrophysiol. 2025 Oct;68(7):1409-1415. doi: 10.1007/s10840-023-01468-1. Epub 2023 Jan 18. PMID 36652082
- See also: manuscript — https://link.springer.com/article/10.1007/s10840-023-01468-1